CLINICAL TRIAL: NCT05703841
Title: An Open-label, Single-dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of JNJ-77242113 Following Oral Administration in Healthy Chinese Adult Participants
Brief Title: A Study of JNJ-77242113 Following Oral Administration in Healthy Chinese Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR109263; 77242113PSO1004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2023-01-20; First posted 2023-01-30 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1: JNJ-77242113 Dose 1 (Experimental): Participants will receive a single oral dose of JNJ-77242113 Dose 1 on Day 1.
  Interventions: Drug: JNJ-77242113
- Cohort 2: JNJ-77242113 Dose 2 (Experimental): Participants will receive a single oral dose of JNJ-77242113 Dose 2 on Day 1.
  Interventions: Drug: JNJ-77242113
- Cohort 3: JNJ-77242113 Dose 3 (Experimental): Participants will receive a single oral dose of JNJ-77242113 Dose 3 on Day 1.
  Interventions: Drug: JNJ-77242113

INTERVENTIONS:
Drug: JNJ-77242113 — JNJ-77242113 will be administered orally as an immediate-release (IR) file-coated tablet.
  Other Names: PN-21235; PN-235

SUMMARY:
The purpose of the study is to assess what drug does to body when healthy Chinese participants receive single oral dose of JNJ-77242113.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening. If there are any abnormalities, they must be consistent with the underlying illness in the study population or considered not clinically relevant and this determination must be recorded in the participant's source documents and initialed by the investigator
* Body mass index (BMI; weight kilograms [kg] per height [meter^2]) between 18.0 and 27.9 kilograms per meter^2 (kg/m2) (inclusive), and body weight not less than 50.0 kg at screening
* A woman of childbearing potential must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) at screening and on Day -1
* Blood pressure (after the participant is supine for 5 minutes) between 90 (inclusive) and 140 millimeters of mercury (mmHg) (exclusive) systolic, and no higher than 90 mm Hg diastolic
* Must be a nonsmoker or habitually smokes no more than 5 cigarettes or equivalent of e-cigarettes, or 2 cigars, or 2 pipes of tobacco per day for at least 6 months before study drug administration

Exclusion Criteria:

* History of surgical resection of the stomach, small or large intestine (excluding appendectomy, cholecystectomy, or resection of benign polyps)
* History of use of medications such as nonsteroidal anti-inflammatory drugs (NSAIDS) or aspirin within 28 days prior to screening or planned use during the study
* Clinically significant infection within 30 days prior to screening or any serious infection within 6 months prior to screening requiring intravenous antimicrobial therapy
* Known allergies, hypersensitivity, or intolerance to JNJ-77242113 or its excipients
* History of severe allergic or anaphylactic reactions

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration versus Time Curve From Time Zero to Time of the Last Measurable Concentration (AUC[0-last]) of JNJ-77242113 | Predose up to Day 3
  AUC(0-last) is defined as area under the plasma concentration versus time curve from time zero to time of the last measurable concentration of JNJ-77242113.
Area Under the Plasma Concentration versus Time Curve From Time Zero to Infinite Time (AUC[0-infinite]) of JNJ-77242113 | Predose up to Day 3
  AUC(0-infinite) is defined as area under the plasma concentration versus time curve from time zero to infinite time of JNJ-77242113.
Maximum Observed Plasma Concentration (Cmax) of JNJ-77242113 | Predose up to Day 3
  Cmax is defined as maximum observed plasma concentration of JNJ-77242113.
Time to Reach the Maximum Observed Plasma Concentration (Tmax) of JNJ-77242113 | Predose up to Day 3
  Tmax is defined as time to reach the maximum observed plasma concentration of JNJ-77242113.
Apparent Elimination Half-life (T1/2) of JNJ-77242113 | Predose up to Day 3
  T1/2 is defined as apparent elimination half-life associated with the terminal slope of the semilogarithmic drug concentration-time curve of JNJ-77242113.
Apparent Total Systemic Clearance (CL/F) of JNJ-77242113 | Predose up to Day 3
  CL/F is defined as apparent total systemic clearance after extravascular administration of JNJ-77242113.
Apparent Volume of Distribution (Vz/F) of JNJ-77242113 | Predose up to Day 3
  Vz/F is defined as apparent volume based on terminal phase after extravascular administration of distribution of JNJ-77242113.

SECONDARY OUTCOMES:
Number of Participants with Abnormalities in Physical Examinations | Up to Day 35
  Number of participants with abnormalities in physical examinations will be reported.
Number of Participants with Abnormalities in 12-Lead Electrocardiogram (ECG) | Up to Day 35
  Number of participants with abnormalities in 12-lead ECGs will be reported.
Number of Participants with Abnormalities in Vital Signs | Up to Day 35
  Number of participants with abnormalities in vital signs (including body temperature, pulse rate, respiratory rate, and blood pressure) will be reported.
Number of Participants with Abnormalities in Clinical Laboratory Tests | Up to Day 35
  Number of participants with abnormalities in clinical laboratory tests (including hematology, clinical chemistry, and urinalysis) will be reported.
Number of Participants with Adverse Events (AEs) | Up to Day 35
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency